CLINICAL TRIAL: NCT06274840
Title: COVID-19 Antibody Responses In Cystic Fibrosis: CAR-CF
Brief Title: COVID-19 Antibody Responses In Cystic Fibrosis
Acronym: CAR-CF
Status: Recruiting | Type: Observational
Sponsor: Pilar Azevedo (Other)
Collaborators: Queen's University, Belfast (Other); European Cystic Fibrosis Society - Clinical Trials Network (Other); Cystic Fibrosis Foundation (Other); Medical University Innsbruck (Other)
Responsible Party: Sponsor-Investigator, Pilar Azevedo, Pilar Azevedo, Centro Hospitalar Universitário Lisboa Norte
Organization: Centro Hospitalar Universitário Lisboa Norte (Other)
Other Study IDs: CAR-CF
Record Dates: First submitted 2024-02-21; First posted 2024-02-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; Cystic Fibrosis
MeSH Terms: conditions — COVID-19; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus disease 2019 (COVID-19) which is caused by the virus SARS-CoV-2 has resulted in an ongoing global pandemic. It is unclear whether the relatively low number of reported cases of COVID-19 in people with CF (pwCF) is due to enhanced infection prevention practices or whether pwCF have protective genetic/immune factors. This study aims to prospectively assess the proportion of pwCF, including both adults and children with CF who have evidence of SARS-CoV-2 antibodies over a two-year period. This study will also examine whether pwCF who have antibodies for SARS-CoV-2 have a different clinical presentation and what impact this has on their CF disease. The proposed study will recruit pwCF from paediatric and adult CF centres in Europe. Serological testing to detect antibodies will be performed on blood samples taken at month 0, 6, 12, 18 and 24 with additional time-points if bloodwork is available via normal clinical care. Clinical data on, lung function, CF-related medical history, pulmonary exacerbations, antibiotic use, and microbiology and vaccination receipt, will be collected during routine clinical assessments.

Associations will be examined between socio-demographic and clinical variables and serologic testing. The effects of SARS-CoV-2 infection on clinical outcomes and analyse end-points will be examined to explore any age-related or gender-based differences, as well as subgroup analysis of outcomes in lung-transplant recipients and pwCF receiving CFTR modulator therapies. As pwCF receive COVID-19 vaccination a comparison of the development and progression of anti-SARS-CoV-2 antibodies in pwCF following natural infection and vaccination SARS-CoV-2 over time will be performed.

DETAILED DESCRIPTION:
This is a prospective, longitudinal cohort study in people with Cystic Fibrosis (pwCF) that involves repeated serial sampling of participants. This study design was chosen to provide comprehensive information on SARS-CoV-2 seroprevalence changes over time and the subsequent clinical impact on pwCF. The study will be conducted at participating CF centres over a 3-year period. Study participants will include paediatric and adult pwCF. Participating investigators can enrol all eligible pwCF over a 12-month period. Participants are then followed up for 24 months. Participants will donate blood samples at their routine clinic visits. Blood samples will be collected at Day 0 (baseline), at Months 6, 12, 18 and 24 (to coincide with routine clinical reviews). Additional blood samples will be taken opportunistically every time the participant visits the clinic for blood draws. These blood samples could be related to, routine care, annual review visits, pulmonary exacerbations (PEx), CF complications or when initiating new treatments (e.g. CFTR modulators).

Serum from blood samples will be shipped to a central laboratory (Queen's University Belfast) for standardized measurement of SARS-CoV-2 antibodies.

Alongside the blood samples the investigators will also collect clinical data from the patient's health records and will input this data into the case report form (CRF). Clinical data will be collected in conjunction with routine care visits, according to local clinical practice. Investigators will collect data elements from information routinely recorded in the patients' medical records. Data will be collected at baseline, month 6, 12, 18 and 24 as per the study schedule, and at additional blood sampling timepoints as previously explained above. Data collection will include routine data available from CF clinic follow-ups including background demographic information, CF medical

history, medications, exacerbation information, sputum microbiology and clinical and lung function parameters. Information on SARS-CoV-2 infection history and vaccine receipt will also be collected.

The maximum follow-up duration of participation in the study for each patient will be 24 months. This study duration (24-month follow-up) is justified as it provides sufficient time to observe changes in antibody prevalence over the course of the COVID-19 pandemic as well as sufficient time to determine long term clinical outcomes for pwCF who are SARS-CoV-2 seropositive. Furthermore, investigators anticipate the 2-year study follow-up period will provide sufficient time to observe the impact of vaccination on antibody levels given that a number of vaccines are now commercially available.

The investigators will compare the level of antibody responses between natural COVID-19 infection and vaccination in pwCF and how this varies over time. This will be achieved by analyzing seroprevalence and antibody levels according to natural infection and vaccination status and according to time of sample post infection or post vaccination, if known.

Optional Study sample collection:

For participants who consent, a second blood sample will also be drawn into EDTA tubes (plasma). Consent to this optional study sample would allow this sample and any remaining serum (following antibody testing) to be stored for future analysis and allow further research to be carried out on related studies to COVID-19 and CF

ELIGIBILITY:
Inclusion Criteria:

* Consenting people with cystic fibrosis of any age, genotype, transplant status and disease severity

Exclusion Criteria:

* Refusal to give informed consent
* Contraindication to venepuncture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consenting people with cystic fibrosis of any age, genotype, transplant status and disease severity will be eligible to participate in the study. The study population is expected to be representative of the general CF population.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
SARS-COV-2 seroprevalence | 3-year period (comprising a 1-year enrollment period and a 2-year follow-up)
  proportion of pwCF with at least 1 seropositive result over the study period and the difference in this proportion by age, geographical area and over time.
Association of SARS-CoV-2 seropositivity, clinical symptoms and clinical outcomes in pwCF | 3-year period (comprising a 1-year enrollment period and a 2-year follow-up)
  incidence of symptomatic COVID-19 over the study period and severity; proportion of seropositive pwCF with subsequent CF exacerbation compared to pwCF who are seronegative; death rate in pwCF with at least one seropositive result compared to pwCF who are seronegative.
Longitudinal comparison of the detection | 3-year period (comprising a 1-year enrollment period and a 2-year follow-up)
  including level and duration of anti-SARS-CoV-2 antibodies in pwCF following natural infection and SARS-CoV-2 vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- CHLN, Lisbon, Portugal